CLINICAL TRIAL: NCT00366522
Title: Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of LXR-623 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating LXR-623 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3201A1-100
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Safety; Healthy; healthy subjects
MeSH Terms: interventions — 2-(2-chloro-4-fluorobenzyl)-3-(4-fluorophenyl)-7-(trifluoromethyl)-2H-indazole

INTERVENTIONS:
Drug: LXR-623

SUMMARY:
To evaluate the safety and tolerability of a single dose of LXR-623 in healthy subjects.

ELIGIBILITY:
Inclusion:

* Healthy, men or women, aged 19-50 years

Exlcusion:

* Use of any investigational or prescription drug within 30 days before study start
* Any clinically imprtant medical disease or abnormal laboratory test results

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Lincoln, Nebraska, United States